CLINICAL TRIAL: NCT00465881
Title: Observational Study of Interstitial Glucose Monitoring With the FreeStyle Navigator Continuous Glucose Monitoring (CGM) System to Develop Novel Methods for Displaying, Reporting and Analyzing CGM Data for Clinical Decision-Making
Brief Title: Develop Novel Methods to Display, Report and Analyze CGM Data for Clinical Decision-Making in People With Diabetes
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Collaborators: Abbott Diabetes Care (Industry)
Other Study IDs: 01929-05-C
Record Dates: First submitted 2007-04-24; First posted 2007-04-25 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2007-09

CONDITIONS: Diabetes; Glucose Variability; CGM
Keywords: Diabetes; CGM
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: CGM System for Type 1 and Type 2 Diabetes Mellitus

SUMMARY:
The purpose of this study is to obtain sufficient continuous glucose monitoring (CGM) data in a manner that provides clinical information that is not available using conventional self-monitored blood glucose. Currently, a formal method does not exist for evaluating CGM data except for looking at each glucose reading across the days a CGM system has been worn and evaluating it based on clinical practice experience. The hope is that a mathematical model can be developed that will enable health care providers to quickly and easily determine what changes in diabetes treatment need to be made after CGM data is obtained.

DETAILED DESCRIPTION:
There are two purposes to the study. First, to use an investigational device, the FreeStyle Navigator Continuous Glucose Monitoring (CGM) System (Abbott Diabetes Care) to obtain sufficient longitudinal data in order to develop a method for reporting CGM data in a manner that provides clinical information that is not available using conventional SMBG. The long-term goad is to determine the manner and degree to which CGM contributes to clinical decision-making. Because of the evidence that glucose regulation may be indirectly related to blood pressure levels, a second purpose of the study is to monitor variation in BP control by means of self-monitored BP.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Diagnosed with type 1 or type 2 diabetes
* Treated with insulin therapy
* Can also be taking other diabetes medication treatment
* Age 21 and older
* Willing to give informed consent
* Capable of following the protocol and instructions of study staff
* Available for scheduled visits
* Access to telephone communications

Exclusion Criteria:

* Under 21 years of age
* Unable to follow protocol
* Unable to read and write in English
* Skin abnormalities at insertion sites
* Allergy to adhesives
* Any concomitant medication thay would likely affect evaluation of device

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-01; Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger S. Mazze, PhD, Principal Investigator — International Diabetes Center - Park Nicollet Institute; Richard M. Bergenstal, MD, Principal Investigator — International Diabetes Center - Park Nicollet Institute; Ellie S. Strock, RN BC-ANP, Principal Investigator — International Diabetes Center - Park Nicollet Institute
Locations (1):
- International Diabetes Center - Park Nicollet Health Services, Minneapolis, Minnesota, United States